CLINICAL TRIAL: NCT01854281
Title: Nitrogen Bubble Detection After Simulated Dives in Divers With PFO and After PFO Closure
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Jakub Honek, MD, MD, University Hospital, Motol
Other Study IDs: EK-1929/12
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Patent Foramen Ovale
Keywords: Patent foramen ovale; Catheter-based closure; Nitrogen bubbles; Decompression sickness
MeSH Terms: conditions — Foramen Ovale, Patent; Decompression Sickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patent foramen ovale dive A group: Divers with a previously diagnosed patent foramen ovale observed after Dive A.
- Closure dive A group: Divers with a patent foramen ovale previously closed by a catheter-based procedure observed after Dive A.
- patent foramen ovale dive B group: Divers with a previously diagnosed patent foramen ovale observed after Dive B.
- closure dive B group: Divers with a patent foramen ovale previously closed by a catheter-based procedure observed after Dive B.

SUMMARY:
The aim of this study is to determine whether catheter-based closure of patent foramen ovale is effective in preventing paradoxical embolization of nitrogen bubbles after simulated dives.

DETAILED DESCRIPTION:
The aim of this study is to determine whether catheter-based closure of patent foramen ovale (PFO) is effective in preventing paradoxical embolization of nitrogen bubbles after simulated dives.

Ultrasonographic detection of venous and arterial nitrogen bubbles will be performed in divers after surfacing from simulated dives in hyperbaric chambers. Divers will be observed after two different dive profiles - Dive A (dive to 18 m for 80 min bottom time) and dive B (dive to 50 m for 20 min bottom time), both performed according to US Navy Air decompression procedure 1996. For both dives two groups will be compared: Divers with PFO and divers after previous catheter-based closure of PFO.

The study will be observational. Sonographic detection of bubbles will be performed after simulated dives that are part of a training program of the divers. Two different dives, previously documented to generate significant amount of venous nitrogen bubbles, were chosen.

The primary end-point will be a positive transcranial doppler test (defined as one or more bubbles detected either during native breathing or after Valsalva maneuver).

Inclusion criteria are: 1) previously diagnosed PFO or a PFO that has been occluded by a catheter-based procedure, 2) signed informed consent

Exclusion criteria: 1) another dive performed in the preceding 24 hours, 2) another previously diagnosed right-to-left shunt, 3) disagreement to be included in the study

This study will be single-center.

ELIGIBILITY:
Inclusion Criteria:

1. previously diagnosed PFO or a PFO that has been occluded by a catheter-based procedure
2. signed informed consent

Exclusion criteria:

1. another dive performed in the preceding 24 hours
2. another previously diagnosed right-to-left shunt
3. disagreement to be included in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult scuba divers with either a previously diagnosed patent foramen ovale (PFO) or after a catheter-based PFO closure. Consecutive divers that undergo a simulated dive in hyperbaric chamber will be recruited.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Veselka, MD, PhD, Study Chair — Department of Cardiology, UH Motol; Jakub Honek, MD, Study Director — Department of cardiology, UH Motol
Locations (1):
- Department of Cardiology, University Hospital Motol, Prague, Czechia

REFERENCES:
- [Derived] Honek J, Sramek M, Sefc L, Januska J, Fiedler J, Horvath M, Tomek A, Novotny S, Honek T, Veselka J. Effect of catheter-based patent foramen ovale closure on the occurrence of arterial bubbles in scuba divers. JACC Cardiovasc Interv. 2014 Apr;7(4):403-8. doi: 10.1016/j.jcin.2013.12.199. Epub 2014 Mar 14. PMID 24630875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were included consecutively in the Hyperbaric chamber of the Regional hospital Kladno, Kladno, Czech Republic and at Hyperbaric chamber Vyškov, Vyškov, Czech Republic, where they performed a training dive. Two dive profiles were performed (dive A and Dive B). The recruitment took part between 15/May/2013 and 15/June/2013.
Pre-assignment Details: No participants were excluded from the study, all enrolled participants completed the study, no transition between groups occured.
Period: Overall Study
Arm/Group | Closure Dive A Group | Patent Foramen Ovale Dive A Group | Closure Dive B Group | Patent Foramen Ovale Dive B Group
Started | 15 | 19 | 5 | 8
Completed | 15 | 19 | 5 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Closure Dive A Group | Patent Foramen Ovale Dive A Group | Closure Dive B Group | Patent Foramen Ovale Dive B Group | Total
Number analyzed (Participants) | 15 | 19 | 5 | 8 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 19 | 5 | 8 | 47
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (8.5) | 33 (7.6) | 33 (12.1) | 33 (4.8) | 35 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 1 | 0 | 9
  Male | 12 | 14 | 4 | 8 | 38
Region of Enrollment [Number; unit: participants]
  Czech Republic | 15 | 19 | 5 | 8 | 47
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 27.3 (3.9) | 25.9 (4.2) | 28.3 (5.7) | 25.2 (2.2) | 26.3 (3.9)
Number of dives [Mean (Standard Deviation); unit: Dives] — Total number of dives in history reported by the diver.
  Dives | 1237 (1762) | 412 (984) | 998 (1851) | 191 (339) | 622 (1238)
Number of decompression dives [Mean (Standard Deviation); unit: Dives] — Total number of decompression dives in history reported by the diver.
  Dives | 251 (314) | 70 (180) | 150 (162) | 44 (82) | 127 (228)
history of decompression sickness [Number; unit: participants] — number of divers with history of decompression sickness as reported by the divers.
  participants | 14 | 10 | 4 | 3 | 31

OUTCOME MEASURES:

1. Primary Outcome: Arterial Nitrogen Bubbles After Surfacing
Description: Arterial gas bubbles are detected by transcranial doppler ultrasonography. Positive outcome is 1 or more bubbles detected.
Time Frame: assesed within 1 hour after surfacing
Measure: Number; unit: participants
Arm/Group | Closure Dive A Group | Patent Foramen Ovale Dive A Group | Closure Dive B Group | Patent Foramen Ovale Dive B Group
Number analyzed (Participants) | 15 | 19 | 5 | 8
participants | 0 | 6 | 0 | 7
Statistical Analysis 1: Comparison: Closure Dive A Group vs Patent Foramen Ovale Dive A Group; null hypothesis: there is no difference in the occurence of arterial bubbles after simulated dive between closure and PFO groups; Test type: Superiority or Other; p = 0.02, Fisher Exact
Statistical Analysis 2: Comparison: Closure Dive B Group vs Patent Foramen Ovale Dive B Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Closure Dive A Group | Patent Foramen Ovale Dive A Group | Closure Dive B Group | Patent Foramen Ovale Dive B Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 0/15 | 4/19 | 0/5 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closure Dive A Group (N=15) | Patent Foramen Ovale Dive A Group (N=19) | Closure Dive B Group (N=5) | Patent Foramen Ovale Dive B Group (N=8)
Mild neurological symptoms of decompression sickness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) — All patients were questioned and examined by physician after the dive. Headache, fatigue, visual problems, paresthesia were considered mild neurological symptoms of decompression sickness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes